CLINICAL TRIAL: NCT06694311
Title: Physiologic Effects of Two Non-invasive Respiratory Support Therapies (continuous Positive Airway Pressure Vs High Flow Nasal Oxygenation) in Patients with Acute Respiratory Distress Syndrome: a Randomized Clinical Trial.
Brief Title: Physiologic Effects of Continuous Positive Airway Pressure and High Flow Nasal Oxygenation in Patients with Acute Respiratory Distress Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ricard Mellado Artigas (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Spanish Society of Pneumology and Thoracic Surgery (Other)
Responsible Party: Sponsor-Investigator, Ricard Mellado Artigas, Senior Specialist, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HCB/2023/1105
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Acute Respiratory Failure with Hypoxia
Keywords: Acute respiratory distress syndrome (ARDS); Continuous positive airway pressure (CPAP); High flow nasal oxygenation; Patient self-inflicted lung injury (P-SILI); Soluble receptor of advanced glycation end-products (sRAGE); Transpulmonary pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: This is a multicentric, randomized, open label, controlled, superiority clinical trial. Participants will undergo permuted block randomization with a ratio 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP (Experimental): CPAP 12 cmH2O
  Interventions: Device: CPAP
- HFNO (Active Comparator): HFNO 50 L/min.
  Interventions: Device: HFNO 50 L/min

INTERVENTIONS:
Device: CPAP — 12 cmH2O for 48 hours (at least 10 hours of therapy per day). Nasobucal interface will be the preferred route with complete facial mask being also an acceptable device. If needed, therapy breaks will be delivered with HFNO at 50 L/min.
  Non-invasive ventilation will not be allowed.
  After 48 hours of treatment, clinicians will be able to decide the respiratory support to be provided although CPAP will be recommended to be continued as long as PaO2/FiO2 is less than or equal to 300 and inspired oxygen fraction is 40% or more.
  Arms: CPAP
Device: HFNO 50 L/min — HFNO 50 L/min for 48 hours. Therapy breaks with oxygen facemask will be allowed as per clinician decision but the protocol will advise against this practice.
  Non-invasive ventilation will not be allowed.
  After 48 hours of treatment, clinicians will be able to decide the respiratory support to be provided although HFNO will be recommended to be continued as long as PaO2/FiO2 is less than or equal to 300 and inspired oxygen fraction is 40% or more.
  Arms: HFNO

SUMMARY:
The acute respiratory distress syndrome (ARDS) consists on a lack of breath due to fluid overload in the lungs that is not produced by a heart desease. Some people with this condition may need to be intubated and connected to invasive mechanical ventilation, but less severe cases may need supplementary oxygen that can be delivered with non-invasive devices, such as CPAP (continuous positive airway pressure) or HFNO (high flow nasal oxygenation). CPAP consists on a facemask that provides oxygen-enriched air at a high pressure, whereas HFNO consists on nasal cannula that provides oxygen-enriched air at a high flow.

Patients with ARDS may present with high respiratory efforts that can eventually damage their own lungs and contribute to the development of a phenomenon known as patient self-inflicted lung injury (P-SILI). Previous research has identified that CPAP may be successful in attuenuating P-SILI compared to HFNO, but it is not known whether this attenuation actually results into a reduction in lung injury in real patients.

In this multicentre trial, 120 non-intubated patients with stablished ARDS will be randomly assigned to receive oxygen-enriched air through either CPAP or HFNO for 48 hours plus standard intensive care. The primary goal of this study is to determine the pulmonary effect of CPAP and HFNO through lung injury biomarkers that can be detected in blood, such as sRAGE (soluble Receptor of Advanced Glycation End-products), angiotensin-II, interleukin-6 and interleukin-10. It will also be studied whether CPAP reduces 48-hour traqueal intubation rate, 90-day traqueal intubation rate and 90-day mortality.

Identifying that CPAP attenuates lung injury in spontaneously breathing ARDS patients will help clinicians to better understand this condition and to better treat this patients, so they do not evenutally need traqueal intubation and connection to invasive mechanical ventilation.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is defined as an acute hypoxemic respiratory failure with non-cardiogenic pulmonary opacities. This condition has been recently extended to non-intubated patients. Patients under non-invasive respiratory support might present with high transpulmonary pressures, pulmonary strain and pendelluft, which contribute to the development of patient self-inflicted lung injury (P-SILI). Previous studies have identified that continuous positive airway pressure (CPAP) is successful in attenuating P-SILI effectors compared to high flow nasal oxygenation (HFNO). However, it remains uncertain whether this attenuation actually results into a reduction in lung injury and improved clinical outcomes.

This is a multicentre, randomised, open-label, controlled trial. 120 non-intubated patients with established ARDS will be randomly assigned to receive non-invasive respiratory support with either CPAP 12 cmH2O or HFNO 50 L/min for 48 hours plus standard intensive care. The primary outcome is biological lung injury evaluated through the epithelial pulmonary dysfunction biomarker sRAGE (soluble Receptor of Advanced Glycation End-products). Secondary outcomes include plasmatic pulmonary dysfunction biomarkers (angiotensin-II, interleukin-6, interleukin-10), P-SILI effectors (pulmonary strain, pendelluft, transpulmonary pressure), 48-hour traqueal intubation rate, 90-day traqueal intubation rate and 90-day mortality. All analyses will be conducted according to the intention-to-treat principle.

This study will assess the potential role of CPAP in attenuating P-SILI effectors and inflicting less biological lung injury compared to HFNO. This physiologic effect may lead to lower rates of traqueal intubation and mortality. This project will provide new knowledge on the respiratory management of non-intubated ARDS patients, a subject where evidence is lacking.

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 ratio <300 mmHg with FiO2 >40% and PEEP ≥5 cmH2O (CPAP) or flow ≥30 L/min (HFNC).
* Bilateral pulmonary opacities observed in the chest X-ray, thoracic computerized tomography (CT) scan or lung ultrasonography (bilateral B lines)
* <7 days from the pulmonary insult to symptom onset and criteria 1 and 2
* Not meeting the aforementioned criteria for >24 hours prior to study inclusion.

Exclusion Criteria:

* Age <18 years or >80 years
* History of chronic respiratory failure or interstitial pulmonary disease
* Acute cardiogenic pulmonary edema after echocardiographic evaluation
* Having received either invasive mechanical ventilation or non-invasive mechanical ventilation (NIV)
* Atelectasis, pleural effusion, pulmonary masses or nodules as the primary finding in thoracic imaging.
* "Do not intubate, do not resuscitate" orders
* Presenting significant nasal obstruction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
sRAGE | From enrollment to the end of treatment at 48 hours.
  The primary outcome of this project is sRAGE, a plasma biomarker indicative of pulmonary epithelial dysfunction. This comparator was selected due to its established association with ventilator-induced lung injury (VILI) and mortality in intubated ARDS patients. sRAGE has got an excellent capacity to detect driving pressure >14 cmH2O in ARDS patients undergoing invasive mechanical ventilation. This suggests that sRAGE may be an adequate biomarker for detecting pulmonary strain in non-intubated ARDS patients.

SECONDARY OUTCOMES:
Angiotensin-II | From enrollment to the end of treatment at 48 hours.
  Endothelial pulmonary injury plasma biomarker.
Interleukin 6 | From enrollment to the end of treatment at 48 hours.
  Systemic inflammation biomarker.
Interleukin 10 | From enrollment to the end of treatment at 48 hours.
  Systemic inflammation biomarker
Orotraqueal intubation | From enrollment to the end of treatment at 48 hours and at 90 days
  Tracheal intubation rate
Mortality | From enrollment to 90 days
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Ferrando Ortolá, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Vallverdu J, Barbeta E, Mellado R, Torres A, Ferrando C. Physiologic effects of two non-invasive respiratory support therapies (continuous positive airway pressure versus high-flow nasal oxygenation) in patients with acute respiratory distress syndrome: study protocol for a randomized clinical trial. Trials. 2026 Jan 2. doi: 10.1186/s13063-025-09344-1. Online ahead of print. PMID 41484920